CLINICAL TRIAL: NCT04700293
Title: Tolerance and Acceptability Evaluation of AYMES AMSTERDAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AY:AMS
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AYMES AMSTERDAM (Experimental): Patients established on an oral nutritional supplement (ONS), requiring nutritional supplementation of at least 300kcal/day will be changed onto an equivalent prescription of AYMES 'AMSTERDAM' for a period of > 7 days.
  Interventions: Dietary Supplement: AYMES AMSTERDAM

INTERVENTIONS:
Dietary Supplement: AYMES AMSTERDAM — AYMES AMSTERDAM is a Food for Special Medical Purposes (FSMP) and must, therefore, be used under medical supervision. It is not designed as a sole source of nutrition.

SUMMARY:
To evaluate tolerance and acceptability of 'AMSTERDAM' in patients requiring supplementary oral nutritional support compared with currently available alternatives.

DETAILED DESCRIPTION:
To evaluate tolerance and acceptability of 'AMSTERDAM' in patients requiring supplementary oral nutritional support compared with currently available alternatives, measuring outcomes of GI effects, Compliance, product preference, convenience etc.

To obtain data to support an ACBS submissions for 'AMSTERDAM' (to allow for prescription in the community at NHS expense).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants.
* ≥ 18 years of age.
* Participants of the intended target group (e.g. MUST score ≥ 1) with an anticipated period of nutritional support ≥ 7 days.
* Patient is able and willing to provide written informed consent.

Exclusion Criteria:

* Participants with medical or dietary contraindication to any feed ingredients.
* Participants requiring sole enteral tube feeding or parenteral nutrition.
* Participants with significant renal (requiring dialysis) or hepatic impairment (e.g. hepatitis.)
* Participants with dysphagia requiring levels 1, 2, 3 or 4 thickened fluids.
* Participants with uncontrolled inflammatory bowel disease or previous bowel resection with ongoing gastrointestinal symptoms.
* Participants for whom the investigator has concerns regarding the ability or willingness of the patient and or carer to comply with protocol requirements.
* Participation in any other studies involving investigational or marketed products concomitantly or within 2 weeks prior to entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Tolerance when consuming AYMES AMSTERDAM | 7 days
  To assess gastro-intestinal tolerance of 'AMSTERDAM' in patients in the community requiring oral nutritional supplementation. Monitoring includes recording the number of any GI complaints via a daily diary.

SECONDARY OUTCOMES:
Acceptability and Palatability of Consuming the Nutritional Supplement: questionnaire | 7 days
  To assess the acceptability of 'AMSTERDAM' in patients in the community requiring oral nutritional supplementation. At the end of the intervention period an acceptability and preference questionnaire will be completed by the patient in order to seek their opinion on the taste, smell, texture and overall liking of the new supplement drink. A 5 point hedonic scale will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- AYMES International Ltd., Haywards Heath, United Kingdom

IPD SHARING:
Plan to Share IPD: No